CLINICAL TRIAL: NCT04521491
Title: A Randomized Controlled Study on the Effect of Postoperative Adjuvant Chemotherapy With FOLFOX4 After Hepatocarcinoma Resection Based on Folate Receptor-positive Circulating Tumor Cells
Brief Title: A Trial of Adjuvant Therapy After Hepatocarcinoma Resection Based on Folate Receptor-positive Circulating Tumor Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, MD, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBHKY2020-01-003
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; adjuvant therapy; FOLFOX4; circulating tumor cells; folate receptor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating | interventions — Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX4 (Experimental): Patients who will receive FOLFOX4 chemotherapy after liver resection
  Interventions: Drug: FOLFOX4(infusional fluorouracil [FU], leucovorin [LV], and oxaliplatin [OXA]).
- placebo (No Intervention): No adjuvant therapy after liver resection

INTERVENTIONS:
Drug: FOLFOX4(infusional fluorouracil [FU], leucovorin [LV], and oxaliplatin [OXA]). — FOLFOX4 (OXA 85 mg/m2 intravenously [IV] on day 1; LV 200 mg/m2 IV from hour 0 to 2 on days 1 and 2; and FU 400 mg/m2 IV bolus at hour 2, then 600 mg/m2 over 22 hours on days 1 and 2, once every 2 weeks.All patients in the treatment group will receive FOLFOX4 at most 12 times beginning from the 4th week after liver resection.
  Arms: FOLFOX4

SUMMARY:
The aim of this study is to analyze the therapeutic effect of postoperative adjuvant chemotherapy with FOLFOX4 after hepatocarcinoma resection based on folate receptor-positive circulating tumor cells. Patients receiving curative resection (R0) were randomized to postoperative FOLFOX4 group and no FOLFOX4 group. The time to recurrence, the overall survival as well as the incidence of complications after therapy was observed to confirm the role of postoperative adjuvant therapy of FOLFOX4.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer death globally. Hepatectomy remains the most widely practiced radical treatment for HCC despite having a high associated recurrence rate, approximately 70% at 5 years after surgery, which often hampers further improvement in survival for these patients. And until now although a lot of different adjuvant therapies had been tried in the clinic, but their role in preventing recurrence remain controversial. As a research of a phase Ⅲ randomize study showed that FOLFOX4 (infusional fluorouracil [FU], leucovorin[LV], and OXA) served as palliative chemotherapy can induce higher overall survival, progression-free survival and response rate comparing to doxorubicin in patients with advanced hepatocellular carcinoma from Asia. The safety data was also acceptable. The chemotherapy of FOLFOX has been accepted by many guidelines and recommended for systematic treatment of advanced HCC. However, the effect of this systemic chemotherapy for recurrent HCC after partial hepatectomy remains to be investigated.

Circulating tumor cells (CTC) have played an important role in early diagnosis of tumors, monitoring of recurrence and metastasis, judgment of patient prognosis, and guidance of postoperative adjuvant treatment. CTC counts can be used to assist diagnosis and evaluation of postoperative prognosis. Previous studies have also shown that folate receptors (FR) are highly expressed in HCC. The detection of circulating tumor cells based on folate receptor (FR+CTC) has been proved to be a sensitive and effective method for detecting CTC.

Patients with HCC who received curative liver resection and with the preoperative FR+CTC level higher than 18.4FU/3mL were randomly assigned 1:1 by the doctors to receive placebo(control group) or FOLFOX4 (treatment group). All patients in the treatment group received FOLFOX4 at most 12 cycles beginning from the 4th week after liver resection. The outcomes of patients were evaluated during the 3-years follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCC who received curative liver resection (R0);
2. Karnofsky Performance Score performance over 60;
3. The functions of the kidney, heart and lung and the blood system are normal and fittable for Licardin therapy;
4. The liver function is of grade A or B in Child-Pugh classification;
5. Patients agreed to collect peripheral blood for detection of CTC at the designated time point;
6. Patients should sign the informed consent of this study.

Exclusion Criteria:

1. If postoperative liver function is Child C, it cannot tolerate chemotherapy;
2. Blood transfusion history within 1 month before enrollment;
3. Severe gastroesophagealvarices with red sign or with variceal hemorrhage before;
4. Malignant or metastatic tumor in other sites in last 5 years;
5. Patients can not be followed-up regularly;
6. Patients participating in other trials or received other treatment previously.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival(RFS) | Up to 2 years
  the time from randomization to documented progression

SECONDARY OUTCOMES:
Time to recurrence (TTR) | Up to 2 years
  the time from randomization to documented progression
Overall survival(OS) | Up to 2 years
  the time from randomization to documented progression

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China